CLINICAL TRIAL: NCT07156890
Title: Surveillance of Respiratory Viruses in Healthcare and Animal Workers in the Netherlands
Brief Title: Surveillance of Respiratory Viruses in Healthcare and Animal Workers
Acronym: SENTINEL
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Corine Geurts van Kessel, Medical microbiologist, Erasmus Medical Center
Other Study IDs: NL-005629
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Viruses
Keywords: healthcare workers; respiratory viruses; pandemic preparedness; virus-specific immunity; surveillance; vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples With DNA — 50ml of whole blood per study visit, 1 throat swab per infection, 1 nasal fluid lining collector (nasosorption) per study visit, 1 nasal brush per study visit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care workers: Hospital staff with and without direct contact to patients (HCW)
- Animal workers: Animal workers with direct contact to animals (AW)

SUMMARY:
Outbreaks with viruses occur continuously, and novel viruses or new variants of existing viruses can surface after a zoonotic event or human-to-human transmission. This project proposal is designed to detect early circulation of (novel) respiratory viruses in both symptomatic and asymptomatic participants, either by direct detection of the virus or changes in local or systemic immunity. Additionally, SENTINEL will provide information on infectivity and (protective) immune responses in viral outbreaks or vaccination campaigns.

DETAILED DESCRIPTION:
A well-designed surveillance study in specific cohorts can serve as an early warning system for (1) the introduction of novel viruses (or variants) in the human population, (2) viral immune escape from pre-existing immunity, or (3) virus evolution into more pathogenic variants. Here, we propose prospective sampling of two sentinel groups with high-risk-of exposure to circulating respiratory viruses for the monitoring of both symptomatic and asymptomatic infections, and immune responses to those infections. Hospital staff (HCW) were shown to be good sentinels for the early detection of respiratory viruses, due to their close contact with patients (or colleagues) with respiratory symptoms. Previous studies in HCW during the COVID-19 pandemic have shown that they are a motivated study population, in which sampling at multiple time-points is feasible if the location is close to work and easily accessible. Other interesting sentinels for respiratory viruses are animal workers (AW), as they are exposed to various animal species and infectious viruses, including respiratory viruses with zoonotic potential. History has shown that most major disease outbreaks were preceded by animal-to-human transmission events that remained undetected until large scale human-to-human transmission occurred. The COVID-19 outbreak is the most recent and devastating example. Similarly, the current extensive transmission of influenza virus H5Nx is of concern and has already spilled over into humans on several occasions. Widespread transmission spillover events to mammals could allow the virus to gain mammalian adaptation. In this prospective SENTINEL study, we propose (self)-sampling of participants (starting just before the 2024 respiratory season), during symptomatic infections to identify and genomically characterize the causative respiratory virus. Follow-up visits will be planned to monitor induced local and systemic immune responses. In addition, we propose periodic sampling of participants to assess changes in local and systemic immune parameters caused by unnoticed/asymptomatic infections with respiratory viruses. Finally, participants will be invited for follow up visits after vaccination against respiratory viruses to monitor vaccine induced responses.

This proposal is unique, as we propose to establish biobanks that include paired samples from the upper respiratory tract and peripheral blood, allowing us to study both local and systemic immunity after infection and/or vaccination. More knowledge on local immunity could be crucial for future vaccine design, and application of vaccines in the respiratory tract. SENTINEL will establish a framework that facilitates early detection of viruses that would otherwise stay under the radar until surfacing due to large scale human-to-human transmission. The rapid genomic characterization and isolation of infectious virus will support rapid development of diagnostic assays, giving a head start in case of (re)emergence of a respiratory virus. Additionally, collecting clinical samples over a prolonged period will yield a valuable biobank of blood samples, respiratory tract samples and viruses, of crucial value for future research and/or (retrospective) analysis of respiratory viruses and immune responses directed against these viruses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Health care workers with or without direct patient contact
* Animal workers with or without direct animal contact

Exclusion Criteria:

* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals working at healthcare facilities or facilities with animals (e.g. farms, bird ringers, or slaughterhouses). We will include an average of 250 participants per year, over a maximum of 5 years. 1,000 participants will be recruited in total for the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Main study endpoint | 60 months
  Identification of circulating respiratory viruses by targeted molecular testing in symptomatic participants
Main study endpoint | 60 months
  Identification of circulating respiratory viruses by metagenomic sequencing in symptomatic participants
Main study endpoint | 60 months
  Identification of circulating respiratory viruses by virus culture in symptomatic participants
Main study endpoint | 60 months
  Longitudinal monitoring of local immune responses, for example by, but not limited to, quantitative, qualitative and/or functional antibody assays (ELISA, VNT, PRNT) to detect changes as a proxy for asymptomatic exposure to respiratory viruses.
Main study endpoint | 60 months
  Longitudinal monitoring of systemic immune responses, for example by, but not limited to, quantitative, qualitative and/or functional antibody assays (ELISA, VNT, PRNT) to detect changes as a proxy for asymptomatic exposure to respiratory viruses.

SECONDARY OUTCOMES:
Secondary study endpoint | 60 months
  Evaluating antibody effector function analyses, detection of virus-specific B-cell and T-cell subset analyses by flow cytometry.
Secondary study endpoint | 60 months
  Document symptoms, disease severity, disease duration and disease burden of respiratory tract infections using questionnaires
Secondary study endpoint | 60 months
  Understand virus spill-over risks between humans and animals by sampling of animal care workers
Secondary study endpoint | 60 months
  Isolate and expand rare and/or new virus (variants) variants from clinical samples by virus culture for biobanking and future research like the development of new assays or preparation of virus stocks for in vivo or in vitro studies.
Secondary study endpoint | 60 months
  Biobanking to enable retrospective analysis, for instance to identify earlier circulation in case of a (re)emerging (new) respiratory virus (variant).

CONTACTS AND LOCATIONS:
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided